CLINICAL TRIAL: NCT03304444
Title: A Pilot Study: A Comparison of Liposomal Bupivacaine to Bupivacaine HCl in Transversus Abdominis Planus Block for Abdominal Gynecologic Surgery
Brief Title: A Comparison of Exparel to Bupivacaine in TAP Block for Abdominal Gynecologic Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abington Memorial Hospital (Other)
Responsible Party: Principal Investigator, Heidi Ching, MD, OBGYN Resident Physician, Abington Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FWA00004123
Record Dates: First submitted 2016-09-13; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Gynecologic Cancer; Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine HCl in TAP block (Active Comparator): When performing a bilateral TAP with Bupivicaine 0.25% and the incision is below the umbilicus: 30 ml of 0.25% bupivacaine is drawn up and given on each side after identification of planes by the anesthesiologist (need 2 vials).
  When performing a bilateral TAP with Bupivicaine 0.25% and the incision extends above the umbilicus: 30 ml of 0.25% bupivacaine is drawn up and given on each side after identification of planes by the anesthesiologist (need 2 vials). A 3rd vial of 30 ml 0.25% bupivacaine will be drawn up and is directly infiltrated into the surgical site (above and below the fascia prior to closure of fascia) extending above the umbilicus by the surgeon.
  Interventions: Drug: Bupivacaine
- Liposomal Bupivicaine in TAP block (Experimental): When performing a bilateral TAP with liposomal bupivacaine and the incision is below the umbilicus: the 20 ml vial of liposomal bupivacaine containing 266 mg, will be diluted with 20 ml of 0.25% bupivacaine (containing 50 mg of bupivacaine) and 20 ml saline (60 ml total). That total volume will be divided into two 30 ml syringes, and each will be used (per side) for the TAP blocks.
  Interventions: Drug: liposomal bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — bupivacaine hydrochloride used in TAP block
  Arms: Bupivacaine HCl in TAP block
Drug: liposomal bupivacaine — liposomal bupivacaine used in TAP block
  Other Names: Exparel
  Arms: Liposomal Bupivicaine in TAP block

SUMMARY:
This study evaluates the comparison between liposomal bupivacaine versus bupivacaine HCl in Transversus Abdominis Plane blocks for gynecologic surgery on the length of stay in the hospital, total narcotic use, and overall complications rates.

DETAILED DESCRIPTION:
The proposed pilot study is evaluating the use of Exparel ™ in an anesthesia protocol for patients undergoing major lower abdominal gynecologic surgery. Exparel ™ is a formulation of liposomal bupivicaine that is reputed to have a much longer duration of action compares to bupivacaine. Exparel™ has been originally demonstrated to be safe and effective in bunionectomy and hemorrhoidectomy. It has recently gained FDA approval for all surgical site infiltration including TAP (Transversus Abdominis Planus block) blocks. Exparel™ has also been studied in other procedures and demonstrated reduction in opioid use and median length of stay (LOS).

Currently, patients on the gynecologic oncology service undergoing major abdominal surgery are receiving a type of regional anesthesia using bupivacaine HCl known as a TAP block as part of an effort to decrease narcotic use post-operatively and decrease hospital length of stay. Bupivacaine has a known eight to twelve hour duration of action, thus addressing immediate post operative pain. As Exparel™ is anticipated to have a longer duration of action, the purpose of this study is to determine if TAP blocks with Exparel™ have an advantage over standard TAP blocks with bupivacaine HCl in reducing length of hospital stay in a randomized controlled trial. Our hypothesis is that TAP blocks with Exparel™ will result in reduced length of stay contributing to significant hospital cost savings. Secondary outcomes include total narcotic use (hypothesized to be reduced) and overall complication rates (hypothesized to remain unchanged). Given there are no published data on the efficacy and safety of using Exparel™ in open gynecologic abdominal surgery, this will be a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing planned exploratory laparotomy
* TAP blocks placed after the laparotomy incision is closed, but before the patient is awake, and placed under ultrasound guidance with correct identification of the correct abdominal plane.
* Consent for TAP block signed by patients preoperatively by anesthesiology

Exclusion Criteria:

* All pregnant patients
* All patients under 18 years of age
* minimally invasive surgery such as laparoscopy or robotic assisted laparoscopy
* medical contraindications to use of bupivacaine or liposomal bupivacaine such as severe hepatic and/or renal disease

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Length of stay post operatively in hospital | through study completion, expected to be approximately 1 year in total
  number of hours patient stays post operatively in hospital

SECONDARY OUTCOMES:
total opioid use post operatively in hospital | through study completion, expected to be approximately 1 year in total
  total opioid use in morphine equivalent that patient uses

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Ching, MD, Principal Investigator — OB GYN Resident
Locations (1):
- Abington Hospital Jefferson Health, Abington, Pennsylvania, United States

DOCUMENTS (3):
  • Statistical Analysis Plan (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT03304444/SAP_000.pdf
  • Study Protocol (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT03304444/Prot_001.pdf
  • Informed Consent Form (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT03304444/ICF_002.pdf